CLINICAL TRIAL: NCT02464332
Title: A Phase 1 Study of BLZ-100 Administered by Intravenous Injection in Subjects With Soft Tissue Sarcoma Undergoing Surgery
Brief Title: Safety Study of BLZ-100 in Adult Subjects With Sarcoma Undergoing Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not enroll any subjects
Sponsor: Blaze Bioscience Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BB-003; 261201400046C-0-0-1 (NIH)
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma, Soft Tissue
Keywords: soft tissue sarcoma; BLZ-100; Tumor Paint
MeSH Terms: conditions — Sarcoma | interventions — tozuleristide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BLZ-100 (Experimental): All participants in the study will receive the investigational drug product BLZ-100.
  In part 1 of the study, two dose levels of BLZ-100 will be evaluated (3 mg and 12 mg) in 6 subjects, with a 2-3 post-dose imaging window.
  In part 2 of the study up to 15 additional subjects will be randomized to one of three imaging interval groups (up to 6 subjects/interval): Early Imaging (within 1 day post-BLZ-100 dose), Intermediate Imaging (2 - 3 days post- BLZ-100 dose), and Late Imaging (4 - 7 days post- BLZ-100 dose).
  Interventions: Drug: BLZ-100

INTERVENTIONS:
Drug: BLZ-100 — All subjects enrolled in the study will receive doses of BLZ-100, an investigational drug for imaging tumors.
  Three different imaging windows will be investigated during the study:
  Early Imaging (imaging occurs within 1 day post-BLZ-100 dose); Intermediate Imaging (imaging occurs within 2-3 days post-BLZ-100 dose); Late Imaging (imaging occurs 4-7 post-BLZ-100 dose)
  All subjects in Part 1 of the study will be imaged in the Intermediate Imaging group. Subjects in Part 2 of the study will be randomized into one of the three imaging groups.
  Other Names: Tumor Paint

SUMMARY:
Many types of cancer are primarily treated with surgery and patient survival is directly related to the extent to which the tumor is able to be removed. It is often difficult for surgeons to distinguish tumor tissue from normal tissue, and failure to surgically remove a cancer-affected lymph node or residual cancer at the surgical margin reduces a patient's chance of survival. Moreover, damage to adjacent normal tissue during surgery can result in significant morbidity. The investigators hypothesize that BLZ-100 will improve surgical outcomes by allowing surgeons to visualize the edges of the tumor and small groups of cancer cells that have spread to other sites in real-time as they operate. This is a safety study to assess the safety of BLZ-100 in patients with soft tissue sarcoma undergoing surgery.

DETAILED DESCRIPTION:
Subjects who provide voluntary written informed consent will be screened for eligibility. Subjects meeting all of the inclusion and none of the exclusion criteria will be eligible to participate.

This is a two part study:

Part 1 - Dose Finding: Subjects will be required to arrive at the phase 1 unit for dosing 2-3 days prior to the planned surgical excision. Two dose levels of BLZ-100 (3 mg and 12 mg) will be evaluated in a total of 6 subjects with a 2-3 day post-dose imaging interval (also defined as the Intermediate Imaging interval).

Part 2 - Imaging Interval Assessment: The BLZ-100 dose to be evaluated in Part 2 will be determined by the Protocol Steering Committee following completion of Part 1. In Part 2, up to 15 additional subjects will be randomized into one of three imaging interval groups (up to 6 subjects per group): Early Imaging (within 1 day post BLZ-100 dose), Intermediate Imaging (2-3 days post BLZ-100 dose), and Late Imaging (4-7 days post BLZ-100 dose). Subjects will be required to arrive at the phase 1 unit for dosing between 1 and 7 days prior to planned surgical excision, depending on which imaging interval they are randomized to.

Following dosing, all subjects will be monitored for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male of female subject aged 18-75 years
2. Diagnosis of soft tissue sarcoma, with scheduled surgical removal for treatment for the disease and completion of chemotherapy or radiation within 4 weeks of BLZ-100 administration
3. Able to provide written informed consent
4. If of child-bearing potential, agree to continued use of two reliable methods of contraceptive from study entry (time of informed consent) through 30 days after BLZ-100 administration
5. Available for all study visits and able to comply with all study requirements

Exclusion Criteria:

1. Clinically-suspected and/or pathologically-confirmed sarcoma of the bone (e.g. osteosarcoma, Ewing's sarcoma with bony involvement, chondrosarcoma, Kaposi's sarcoma, extraosseous primitive neuroectodermal tumor [PNET])
2. Evidence of metastatic disease
3. Female who is lactating/breastfeeding
4. Female with a positive pregnancy test or who is planning to become pregnant during the duration of the study
5. Karnofsky Performance Status of <60%
6. Any of the following laboratory abnormalities at Screening:

   * Neutrophil count <1.5 x 10^9/L
   * Platelets <75 x 10^9/L
   * Hemoglobin <10 g/dL (may be determined following transfusion)
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3x upper limit of normal (ULN)
   * Total bilirubin >1.5x upper limit of reference range (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction)
   * Internal Normalized Ratio (INR) >1.5
   * Creatinine >1.5x ULN
   * Calculated estimated glomerular filtration rate (eGFR) ≤60 mL/min
7. Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV)
8. QTc prolongation >450 msec
9. History of hypersensitivity or allergic reactions requiring corticosteroids, epinephrine, and/or hospitalization
10. Uncontrolled asthma or asthma requiring oral corticosteroids
11. Known or suspected sensitivity to imaging agents that may be used in clinical assessment of this study
12. Known or suspected sensitivity to indocyanine green (ICG)
13. Unstable angina, myocardial infarction, known or suspected transient ischemic events, or stroke within 24 weeks of start of Screening
14. Uncontrolled hypertension
15. Initiation of new photosensitizing drugs within 30 days of Screening
16. Use of any ongoing medications, which might generate fluorescence or, according to the medication label, might generate a photochemical reaction. These include haematoporphyrin derivatives and purified fractions, Photofrin®, and the precursors of protoporphyrin IX (5-Aminolevulinic acid) used in Gliolan or Hexvix
17. Receipt of an investigational drug or device within 30 days of enrollment
18. Prior administration of BLZ-100
19. Any concurrent condition, including psychological and social situations, which, in the opinion of the investigator, would adversely impact the subject or the interpretation of the study data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Seven days after study drug administration
  Safety will be assessed by physical examination and measurement of vital signs and laboratory safety parameters.

SECONDARY OUTCOMES:
Change of concentration of BLZ-100 in the blood | Prior to dosing and at 1 minute, 5 minutes, 15 minutes, 30 minutes, 60 minutes and 120 minutes after end of injection, and pre-surgery and 24 hours post-surgery
  BLZ-100 levels in blood will be analyzed by chemical means and these data will be used to calculate pharmacokinetic parameters.
Fluorescence signal from areas of tumor and non-tumor | 1 day post-dose, 2-3 days post-dose, or 3-7 days post-dose
  Fluorescent signal in sections of excised tumor and adjacent normal tissue will be measured using an infrared imaging system.
Ideal combination of dose and imaging interval | 1 day post-dose, 2-3 days post-dose, 3-7 days post-dose
  Fluorescent signal will be evaluated in sections of excised tumor and adjacent normal tissue to determine which imaging interval provides the optimal images.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Forscher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States